CLINICAL TRIAL: NCT00251121
Title: Mini-invasive Electrophysiology Study as a Routine Examination for Patients Complaining of Tachycardia, But With a Negative Holter ECG.
Brief Title: Routine Mini-invasive Electrophysiology Study for Patients Feeling Tachycardia, With a Negative Holter ECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jan Hysing MD PhD, MD. Cardiologist, medical Department Sykehuset i Telemark, Sykehuset Telemark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-05116
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-02

CONDITIONS: Pre-excitation Syndromes; Paroxysmal Tachycardia; Atrial Fibrillation; Atrial Flutter; Wolff-Parkinson-White Syndrome
Keywords: Electrophysiological study; paroxysmal tachycardia
MeSH Terms: conditions — Pre-Excitation Syndromes; Tachycardia, Paroxysmal; Atrial Fibrillation; Atrial Flutter; Wolff-Parkinson-White Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atrial pacing (Experimental): Diagnostic pacing in right heart atrium in order to unmask reentry tachycardia
  Interventions: Other: Mini-invasive electrophysiological study; Other: Atrial pacing

INTERVENTIONS:
Other: Mini-invasive electrophysiological study — Transvenous pacing in right heart atrium
Other: Atrial pacing — Diagnostic pacing in right heart atrium in order to unmask reentry tachycardia

SUMMARY:
Patients complaining of tachycardia but with a negative Holter ECG, are for a limited time period offered a simplified electrophysiological(EP) examination. By a full electrophysiological study(EP study)electrodes are introduced for pacing and sensing i all four heart chambers. Where as by the mini invasive EP study only one electrode is introduced to the right atrium. The simplified procedure represent a smaller risk of complications, requires less resources but should yield the same diagnoses in more than 90% of the cases. The study is a feasibility study to see if the procedure can discover arrythmias in a fairly unselected patient population.

DETAILED DESCRIPTION:
Sykehuset Telemark performs every year approximately 800 Holter ECG examinations. Approximately 200 of these are on the indications tachycardia, and in about 170 patients the examination does not discover any tachycardia Patients who were examined in the period from August 1. 2004 to November 1. 2005 with a negative Holter are mailed a letter with information of the min invasive electrophysiological examination, and an offer of volunteer participation. Patients given their informed consent are then according to waiting list called for the mini-invasive EP-study.

The protocol of the EP stimulation consists of: determination of pacing threshold, pacing with 8 asynchronous beats 600ms and an extrasystole with decremental intervals from 550 ms to 200 ms. The seri is repeated with pacing on 400ms and with two extrasystoles as well as with isoprenaline stimulation.

ELIGIBILITY:
Inclusion Criteria:

* History of complains of tachycardia
* No arrythmias detected by a 24 hours Holter ECG
* Age 19 to 74 years

Exclusion Criteria:

* Patients younger than 18 years
* Patients older than 75

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of tachycardia diagnoses previously not known. | October 2005 to May 2006
  A simple electrophysiologic examination uncovered reentry tachycardia in nine patients and paroxystic atrial flutter in three patients. A total of 56 electrophysiologic examinations were performed, uncovering 12 cases of tachycardia suitable for ablation. Two patients had to undergo DC-conversion, no other complication was observed.
  Interpretation. A simplified electrophysiologic examination of this group of patients will uncover tachycardia suitable for ablation in approximately 20 % of the patients, and increase diagnostic yield of supraventricular tachycardia by 64 %.
Primary outcome was the diagnosis of supraventricular tachycardia suitable for ablation | Oct 2005 - May 2006
  Two patients had to undergo DC conversion for A.fib

SECONDARY OUTCOMES:
Quality of diagnoses after referral to university ref. centre | May 2006 - June 2007
  8 patienst were RF abladed in Oslo University Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hysing, MD. PhD., Principal Investigator — Cardiologist at Medical Department Sykehuset Telemark
Locations (1):
- Sykehuset Telemark, Skien, Telemark, Norway